CLINICAL TRIAL: NCT04101929
Title: A Phase II, Single-arm Study to Evaluate The Safety and Efficacy of Apatinib Combined With Irinotecan and S-1 (ApaIRIS) in Treating Patients With Metastatic Pancreatic Cancer After Chemotherapy With Albumin-bound Paclitaxel Plus Gemcitabine Regimen
Brief Title: Apatinib, Irinotecan and S-1 (ApaIRIS) in Treating Patients With Metastatic Pancreatic Cancer After AG Regimen
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xian-Jun Yu, Prinicipal Investigator, Clinical Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSPAC-25
Record Dates: First submitted 2019-09-22; First posted 2019-09-24 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-11

CONDITIONS: Metastatic Pancreatic Cancer
Keywords: metastatic pancreatic cancer; pancreatic adenocarcinoma; apatinib; S-1; irinotecan
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — apatinib; S 1 (combination); Irinotecan

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Apatinib + S-1+ Irinotecan (Experimental): Apatinib: 250mg po qd； S-1 capsule: According to the body surface area <1.25m2 60mg/d, 1.25 ~ 1.5 m2 80 mg/d, > 1.5m2 100mg/d po bid, taking 7 days, stopping for 7 days, 28 days for 1 cycle; Irinotecan: According to the body surface area of 180 mg/m2, ivgg/90min, once every two weeks.
  Interventions: Drug: Apatinib; Drug: S-1 capsule; Drug: Irinotecan

INTERVENTIONS:
Drug: Apatinib — Patients receive Apatinib 250mg po qd , Treatment repeats every 4 weeks until the disease recurrence or unacceptable toxicity，death or begin a novel therapeutic.
Drug: S-1 capsule — Patients receive S-1 capsule According to the body surface area <1.25m2 60mg/d, 1.25 ~ 1.5 m2 80 mg/d, > 1.5m2 100mg/d po bid, taking 7 days, stopping for 7 days, 28 days for 1 cycle, Treatment repeats until the disease recurrence or unacceptable toxicity，death or begin a novel therapeutic.
Drug: Irinotecan — Patients receive Irinotecan According to the body surface area of 180 mg/m2, ivgg/90min, once every two weeks. Continuous chemotherapy until the criteria for discontinuation of the drug are met (eg, progression of the disease, intolerance of adverse reactions, or withdrawal of informed consent by the patient).
  Because the toxicity of apatinib or irinotecan or tigeol in the chemotherapy regimen meets the withdrawal criteria, the drug can be discontinued alone and the exact duration of the trial treatment recorded.

SUMMARY:
This is a single arm, open label Phase II clinical trial to evaluate the efficacy and safety of apatinib combined with irinotecan and S-1 (ApaIRIS) in treating Patients with metastatic pancreatic cancer after chemotherapy with albumin-bound paclitaxel plus gemcitabine regimen

DETAILED DESCRIPTION:
While AG (albumin-bound paclitaxel + gemcitabine) is one of the preferred first-line chemotherapy for metastatic pancreatic cancer, we have to investigate possible therapeutic options after AG regimen. In this single arm, open-label clinical trial, metastatic pancreatic cancer patients will be received apatinib, irinotecan and S-1. Treatment repeats every 4 weeks until the disease recurrence or unacceptable toxicity, death or begin a novel therapeutic.

The efficacy and safety data will be assessed through PFS, OS, ORR and adverse effects as graded by CTC-AE 5.0.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent and willing to complete the study according to the protocol
* ECOG performance scale ≤ 2;
* Diagnosed as pancreatic adenocarcinoma by histology and cytology;
* Treatment of patients with advanced metastatic pancreatic cancer who have failed with AG (albumin and gemcitabine) regimen
* Baseline blood routine and biochemical indexes meet the following criteria:

  1. Blood routine examination criteria must be met: (no blood transfusion within 14 days)

     1. HB≥90g/L；
     2. ANC≥1.5×109/L；
     3. PLT≥80×109/L
  2. Biochemical tests are subject to the following criteria:

     1. BIL <1.25xULN ；
     2. ALT and AST<2.5ULN；
     3. Serum creatinine. Less than 1 times the upper limit of normal value, Endogenous creatinine clearance>50ml/min ( Cockcroft-Gault formula).
* The advanced pancreatic cancer pathology, with measurable lesions (spiral CT scan is more than 10 mm, according to the standard of RECIST 1.1);
* Life expectancy ≥ 12 weeks;
* Doctors believe that treatment can bring benefits to patients.

Exclusion Criteria:

* unwilling or unable to comply with the study protocol;
* Other or malignant tumors in the past or at the same time, except for cured skin basal cell carcinoma and cervical carcinoma in situ;
* Allergy to apatinib, S-1 raw materials and/or their excipients;
* Received VEGFR inhibitors, such as sorafenib, chougny for treatment;
* Have high blood pressure and antihypertensive drug treatment can not drop to normal range(systolic pressure >140 mmHg, diastolic blood pressure 90>mmHg);
* Suffering from coronary artery disease above grade I, grade I arrhythmia (including corrected QT interval prolongation male > 450 ms, women > 470 MS) and grade I heart insufficiency; urine protein positive patients.
* Renal insufficiency, patients with previous kidney disease, urine protein positive (urinary protein detection 2+ or above, or 24-hour urine protein quantitation > 1.0g);
* Has a variety of factors influencing oral drugs (such as unable to swallow, nausea, vomiting, chronic diarrhea and intestinal obstruction, etc.)
* Pregnant or lactating women;
* Coagulant function abnormality (INR>1.5、APTT>1.5 ULN) with bleeding tendency; Those with bleeding tendency (such as active ulcerative lesions in the stomach, fecal occult blood (++), vaginal and/or hematemesis within 3 months, hemoptysis) or lesions close to the large vessel site;
* Patients with a deficiency of dihydropyrimidine dehydrogenase are known;
* Evidence of any severe or uncontrolled systemic disease (eg, unstable or decompensated breathing, heart, liver or kidney disease, HIV infection, high blood pressure, severe arrhythmia, diabetes, massive active bleeding);
* Patients with a history of psychotropic substance abuse who are unable to quit or have a mental disorder;
* According to the investigator's judgment, there are other serious patients who are at risk to the patient's safety or affect the patient's accompanying disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | through study completion, an average of 1 year
  To investigate the progression-free survival (PFS) of patients with advanced metastatic pancreatic cancer who have failed with AG (albumin and gemcitabine) regimen after treatment with Apatinib combined with Irinotecan and S-1 (ApaIRIS)

SECONDARY OUTCOMES:
Overall Survival | through study completion, an average of 1 year
  To evaluate the overall survival of patients with advanced metastatic pancreatic cancer who have failed with AG (albumin and gemcitabine) regimen after treatment with Apatinib combined with Irinotecan and S-1 (ApaIRIS).
Incidence of Adverse Events | through study completion, an average of 1 year
  Adverse events of patients with advanced metastatic pancreatic cancer who have failed with AG (albumin and gemcitabine) regimen after treatment with Apatinib combined with Irinotecan and S-1 (ApaIRIS).
Overall Response Rate | through study completion, an average of 1 year
  To evaluate the overall response rate of patients with advanced metastatic pancreatic cancer who have failed with AG (albumin and gemcitabine) regimen after treatment with Apatinib combined with Irinotecan and S-1 (ApaIRIS)

CONTACTS AND LOCATIONS:
Overall Officials: Xian-Jun Yu, Study Director — Fudan University
Locations (1):
- Department of Pancreatic and Hepatobiliary Surgery, Fudan University Shanghai Cancer Center; Pancreatic Cancer Institute, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No